CLINICAL TRIAL: NCT04231045
Title: The Impact of Systemic pH on Cardiac Function and Clinical Outcome in the Critically Ill Patient
Brief Title: The Impact of the pH on Cardiac Function in the Critically Ill Patient
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 227870
Record Dates: First submitted 2018-06-22; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Acidosis; Cardiac; Deficiency; Acid Base Disorder
Keywords: acidosis; cardiac contractility; acid-base disorder
MeSH Terms: conditions — Acidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients on PiCCO monitoring system: ALL intensive care patients on PiCCO monitoring system and over 18 years old and on PiCCO for more than 24 hours. Those medical or surgical patients admitted in a UK NHS unit, elective, semi-elective or emergency admission.
  Interventions: Device: PiCCO device cardiac monitoring

INTERVENTIONS:
Device: PiCCO device cardiac monitoring — PiCCO is a cardiac output monitor that combines pulse contour analysis and transpulmonary thermodilution technique.Haemodynamic monitoring
  especially if complex mixed forms of shock (e.g. septic and cardiogenic) PAC unavailable or contra-indicated

SUMMARY:
Study Title: The Impact of the pH on cardiac function in the critically ill patient Sponsor: King's College Hospital NHS Foundation Trust Chief Investigator: Dr Sancho Rodríguez-Villar IRAS Number: 227870

Hypothesis:

Titration studies in animals with normal cardiac function show that a reduction in blood pH (and presumably that of the intracellular and interstitial compartments) from the normal level of 7.40 to 7.20 is associated with a rise in cardiac output. However, when blood pH is less than 7.20, cardiac output is reduced. Similar studies in humans with or without normal cardiac function have not been done, and yet blood pH at which aggressive treatment is recommended has been set at 7.20 based solely on animal experiments. The investigators hypothesize that a change in blood pH in humans will also affect cardiac function, but the level of blood pH at which this is observed might be similar or different in humans. In addition, the presence or absence of underlying cardiac disease and the type of acid-base abnormality present might modify the response of the heart to changes in blood pH.

Primary Objectives:

1. Assess whether there are significant changes in cardiac function associated with changes in blood pH.
2. Relate the changes in cardiac function to the presence or absence of underlying cardiac disease.

Study Design:

A prospective multicenter observational study in 6 ICU´s (between two Trusts). During a year study period, a minimum of 300 patients will be recruited.

DETAILED DESCRIPTION:
Aim The aim of this study is to test the hypothesis that a change in the acidity of the blood (pH) will affect cardiac function in critically ill patients. It will also explore if the presence or absence of underlying cardiac disease and the type of pH abnormality may affect the response of the heart to changes in pH.

Justification for design Blood pH and cardiac function are monitored routinely in critically ill patients and so a prospective observational study design would be a feasible and useful method to address this question.

Inclusion/exclusion criteria explanation In intensive care practice, if a patient requires close cardiac function monitoring clinicians will use a special system for continuously monitoring the cardiac output and other heart functions to guide therapy. The system most commonly used is called PiCCO (pulse contour cardiac output).

Adult patients who are on PiCCO as part of their routine care in ICU for more than 24 hours will be eligible for inclusion in the study.

All patients who do not already have PiCCO in situ will be excluded from the study.

Identification of patients The direct care team will identify all eligible patients in the participating Units. The investigators have agreed to conduct the study in 6 different intensive care units across 2 Trusts and 4 sites - King's College Hospital Foundation Trust - including 3 ICU's at Denmark Hill site and 1 at Princess Royal University Hospital site; Lewisham and Greenwich NHS Trust - including ICU at University Hospital Lewisham and Queen Elizabeth Hospital, Woolwich.

Justification for sample size

In order to examine the relationship between a change in pH and cardiac contractility with power 80% and a 95% confidence interval, it has been calculated that it will be necessary to analyse 363 cases. Statistical analysis will be based on a retrospective audit of the numbers of a patient who fit the criteria, the investigators have assessed that across the 7 units the target sample size will be easily achieved in less than 1 year.

Data collection Data will be collected from ICU charts, medical notes and electronic patient records. This data is routinely collected as part of standard hospital care. The data will be collected by the direct care team and anonymised before it is transferred securely to a statistician for statistical analysis. The patient will not undergo any additional assessments or tests.

Consent All the data to be analysed is routinely collected as part of standard hospital care. There will be no additional tests or assessments in relation to this study. All data will be anonymised prior to analysis therefore, the investigators request approval to enrol patients without obtaining consent.

Data handling A case report form will be completed for each participant. Each participant will be given a unique study identification number. The patient's hospital number will be recorded on the case report form, and data will be collected by the direct care team. When data collection is completed at day 30, the direct care team will remove the top section of the case report form so that the hospital number is removed.

An enrolment log will be stored in the Site File securely on-site in a locked cupboard.

The data will be analysed according to the statistical plan. Results will be published in a peer-review journal.

ELIGIBILITY:
Inclusion Criteria (the three criteria):

* Inclusion Criteria ALL patients on PiCCO monitoring system
* Over 18 years old.
* On PiCCO for more than 24 hours

Exclusion Criteria:

ALL patients WITHOUT PiCCO monitoring system AND:

* < 18 years old
* Vulnerable patients
* Atrial or ventricular arrhythmia: you need a stable pulse to measure the contour.
* Aortic, mitral or tricuspid valve insufficiency. In the case of valve insufficiency the valve does not close correctly. Therefore, the thermodilution curve is affected by indicator regurgitation, resulting in a prolonged indicator decay time.
* Intra-Aortic Balloon pump: once again, the pulse contour is all wrong; but you can still get thermodilution cardiac output measurements.
* Aortic aneurysm: the contour will be bizarre because the arterial compliance is going to be weird, with the aortic aneurysm acting as a damping system by absorbing all the pressure wave.
* Extracorporeal circuit: when you are on bypass, there is no real arterial waveform
* Pneumonectomy: PiCCO relies on there being a relatively normal pulmonary vasculature.
* Massive pulmonary embolism: as above; it is essentially a pneumonectomy by embolism.
* Intracardiac shunt: the PA catheter will also give an inaccurate thermodilution reading.
* Less than a minimal tidal volume 6-8mL/kg
* NON-positive pressure ventilated patients:
* Why does Stroke Volume Variation only apply to positive pressure ventilated patients? It still applies in spontaneously breathing patients; however it is a poorer predictor of fluid responsiveness.
* Why? The sensitivity is decreased: its only 63%. The spontaneous breathing efforts draw a smaller tidal volume, and from such minor changes in thoracic pressure there would insufficient change in ventricle loading; so there may still be changes to stroke volume, but they would be tiny and difficult to measure.
* If there is profound hypovolemia, the IVC can collapse on inspiration. Obviously this decreases preload and confuses your SVV. You cannot predict fluid responsiveness this way, because you never get an accurate impression of preload.
* In spontaneous respiration, inspiration increases the right ventricular preload, which means the right ventricular filling is likely still appeared adequate even if there is some hypovolemia. In spite of low overall volume, the right ventricular preload remains adequate, and thus at least one of the ventricles is likely to be operating in the preload-independent straight part of the Frank-Starling curve
* Severe obesity: In obese patients, Extravascular Lung Water Index (EVLWI) is underestimated because it is related to body weight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UK NHS (National Health service) patients admitted to ICU over 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Assess whether there are significant changes in stroke volume index associated with changes in blood pH using PiCCO technology monitoring. | within 24 hours of being started on the PICCO monitoring system through cardiovascular monitoring study completion, an average of 5 days per patient
  SVI- Stroke Volumen Index (40-60 mL/ m2)
Assess whether there are significant changes in CI -Cardiac index or PCCI are associated with changes in blood pH using PiCCO technology monitoring. | within 24 hours of being started on the PICCO monitoring system through cardiovascular monitoring study completion, an average of 5 days per patient
  CI (Cardiac index or PCCI): 3-5 L/min/m2
Assess whether there are significant changes in CO-Cardiac Output or PCCO are associated with changes in blood pH using PiCCO technology monitoring. | within 24 hours of being started on the PICCO monitoring system through cardiovascular monitoring study completion, an average of 5 days per patient
  CO (Cardiac Output or PCCO): 4 - 8 L/min

SECONDARY OUTCOMES:
Assess whether there are significant changes in cardiac contractility measuring the GEF (Global ejection fraction) are associated with changes in blood pH using PiCCO technology monitoring. | within 24 hours of being started on the PICCO monitoring system through cardiovascular monitoring study completion, an average of 5 days per patient
  GEF (Global ejection fraction): 25- 35% : GEF = (4 x SV) / GEDV. A % of total blood expelled from the heart every beat to the total amount of blood estimated to be present just prior to ventricular systole.
Assess whether there are significant changes in cardiac contractility measuring the dPmx (Index of Left Ventricular Contractility) are associated with changes in blood pH using PiCCO technology monitoring. | within 24 hours of being started on the PICCO monitoring system through cardiovascular monitoring study completion, an average of 5 days per patient
  (dPmx) Index of Left Ventricular Contractility. dPmx is a direct measurement of contractility. The dPmx is a measure of how fast the pressure rises during systole. 900-1200 mmHg/s.
Assess whether there are significant changes in cardiac contractility measuring the CFI (Cardiac function index) are associated with changes in blood pH using PiCCO technology monitoring. | within 24 hours of being started on the PICCO monitoring system through cardiovascular monitoring study completion, an average of 5 days per patient
  CFI (Cardiac function index): 4.5- 6.5 L/min The ratio of the index of cardiac output to the index of the GEDV. A measure of how well the CO is doing in relation to its preload.
Assess whether there are significant changes in cardiac contractility measuring the CPI (Cardiac Power Index) are associated with changes in blood pH using PiCCO technology monitoring. | within 24 hours of being started on the PICCO monitoring system through cardiovascular monitoring study completion, an average of 5 days per patient
  CPI (Cardiac Power Index). Represents the power of left ventricular cardiac output in watts. 0.5-0.7 W/m2

OTHER OUTCOMES:
Assess whether there are significant changes in the preload measuring the ITBVI (Intra thoracic blood volume index) are associated with changes in CO-Cardiac Output PCCO or blood pH using PiCCO technology monitoring. | within 24 hours of being started on the PICCO monitoring system through cardiovascular monitoring study completion, an average of 5 days per patient
  ITBVI(Intra thoracic blood volume index): 850-1000ml/m₂. If not available : ITBVI= GEDI X 1.25
Assess whether there are significant changes in the preload measuring the GEDI (Global end-diastolic volume index) are associated with changes in CO-Cardiac Output PCCO or blood pH using PiCCO technology monitoring. | within 24 hours of being started on the PICCO monitoring system through cardiovascular monitoring study completion, an average of 5 days per patient
  GEDI (Global end-diastolic volume index) 680- 800 mL/m₂

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Lewisham and Greenwhich NHS Trust Foundation, London
  - King´s College Hospital NHS Trust, London

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT04231045/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT04231045/ICF_001.pdf